CLINICAL TRIAL: NCT06694090
Title: Von Willebrand Factor Levels in Patients With Liver Cirrhosis and Portal Hypertension
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Sameh Jakoub Bakhet, Resident doctor, Assiut University
Other Study IDs: Von willebrand factor levels
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Liver Cirrhosis; Portal Hypertension
Keywords: Von willebrand factor; Liver cirrhosis; Portal hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Verify Von willebrand factor role in patients with liver cirrhosis and portal hypertension

DETAILED DESCRIPTION:
Patients with cirrhosis have an endotoxemic medium due to intestinal flora changes, decreased hepatic clearance of endotoxins and transition of bacteria to mesenteric lymph nodes from intestinal barrier .Serum Von Willebrand factor (vWF) increases in a linear ratio with the intensity of endotoxemia.

Portal hypertension (PH) is a hallmark of advanced chronic liver disease (ACLD) that significantly influences the onset of liver-related complications and mortality. It can be quantified using the minimally invasive measurement of the hepatic venous pressure gradient (HVPG). Experimental research has demonstrated that ongoing dysfunction of liver sinusoidal endothelial cells (LSEC) triggers the activation of hepatic stellate cells (HSC) and leads to intrahepatic vasoconstriction, thereby contributing to PH.

Von Willebrand factor (VWF) is released by activated endothelial cells and plays a crucial role in hemostasis by facilitating the adhesion of platelets to subendothelial collagen and other platelet-adhesive proteins exposed during vascular injury. Early studies revealed that VWF levels are elevated in patients with ACLD, linking this finding to endothelial dysfunction likely caused by endotoxemia , resulting from pathological bacterial translocation. Notably, VWF antigen (VWF-Ag) has shown diagnostic potential for clinically significant PH (CSPH; defined by an HVPG ≥ 10 mmHg) and prognostic value for disease progression, even after the underlying cause has been treated.

Elevated VWF levels may help balance the fragile hemostatic system in patients with ACLD by compensating for platelet deficiencies in number and possibly function.

VWF is more than just a hemostatic protein; it serves as a marker of endothelial dysfunction in patients with cirrhosis.VWF levels can independently predict decompensation and mortality in cirrhosis patients, regardless of the stage of liver disease and severity of portal hypertension. The VWF-to-thrombocyte ratio (VITRO) score enhances the diagnostic capability of VWF alone in noninvasively detecting CSPH.In addition to predicting the risk of hepatocellular carcinoma (HCC) in cirrhosis patients, VWF levels also forecast the risk of complications following HCC resection and response to systemic therapies.

ELIGIBILITY:
Inclusion Criteria:

* adult patient >18 years
* both sex male and female
* all stages of liver cirrhosis (compensated and decompensated)

Exclusion Criteria:

* acute liver disease
* any hereditary or acquired diseases that affect VWF level.
* sepsis and infections (including spontaneous bacterial peritonitis), patients with any infectious symptoms at the time of study (increasing VWF Ag levels).
* active extrahepatic malignancies.
* previous liver transplantation.
* any medication affect VWF level.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients aged 18-65 years with all stages of liver cirrhosis (compensated and decompensated)
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Verify Von willebrand factor role in patients with liver cirrhosis and portal hypertension by using VWF-Ag concentation and fibroscan | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kerolos A Sameh, Resident, Principal Investigator — Assiut University; Mohamed A Ramadan, Lecturer, Study Director — Assiut University; Abdelhamid A Mohamed, Lecturer, Study Director — Assiut University

REFERENCES:
- [Result] Foucher J, Chanteloup E, Vergniol J, Castera L, Le Bail B, Adhoute X, Bertet J, Couzigou P, de Ledinghen V. Diagnosis of cirrhosis by transient elastography (FibroScan): a prospective study. Gut. 2006 Mar;55(3):403-8. doi: 10.1136/gut.2005.069153. Epub 2005 Jul 14. PMID 16020491
- [Result] Curakova Ristovska E, Genadieva-Dimitrova M, Caloska-Ivanova V, Misevski J. Von-Willebrand factor as a predictor of three-month mortality in patients with liver cirrhosis compared to MELD score. Acta Gastroenterol Belg. 2019 Oct-Dec;82(4):487-493. PMID 31950803
- [Result] Hametner S, Ferlitsch A, Ferlitsch M, Etschmaier A, Schofl R, Ziachehabi A, Maieron A. The VITRO Score (Von Willebrand Factor Antigen/Thrombocyte Ratio) as a New Marker for Clinically Significant Portal Hypertension in Comparison to Other Non-Invasive Parameters of Fibrosis Including ELF Test. PLoS One. 2016 Feb 19;11(2):e0149230. doi: 10.1371/journal.pone.0149230. eCollection 2016. PMID 26895398
- [Result] van den Boom BP, Stamouli M, Timon J, Bernal W, Blasi A, Adelmeijer J, Fernandez J, Lisman T, Patel VC. Von Willebrand factor is an independent predictor of short-term mortality in acutely ill patients with cirrhosis. Liver Int. 2023 Dec;43(12):2752-2761. doi: 10.1111/liv.15728. Epub 2023 Sep 16. PMID 37715606
- [Result] Elhence A, Shalimar. Von Willebrand Factor as a Biomarker for Liver Disease - An Update. J Clin Exp Hepatol. 2023 Nov-Dec;13(6):1047-1060. doi: 10.1016/j.jceh.2023.05.016. Epub 2023 Jun 2. PMID 37975050
- [Result] Lisman T, Bongers TN, Adelmeijer J, Janssen HL, de Maat MP, de Groot PG, Leebeek FW. Elevated levels of von Willebrand Factor in cirrhosis support platelet adhesion despite reduced functional capacity. Hepatology. 2006 Jul;44(1):53-61. doi: 10.1002/hep.21231. PMID 16799972
- [Result] Pomej K, Scheiner B, Balcar L, Nussbaumer RJ, Weinzierl J, Paternostro R, Simbrunner B, Bauer D, Pereyra D, Starlinger P, Stattermayer AF, Pinter M, Trauner M, Quehenberger P, Reiberger T, Mandorfer M. Clinical significance of substantially elevated von Willebrand factor antigen levels in patients with advanced chronic liver disease. Dig Liver Dis. 2022 Oct;54(10):1376-1384. doi: 10.1016/j.dld.2022.06.010. Epub 2022 Jul 22. PMID 35871985
- [Result] Mandorfer M, Schwabl P, Paternostro R, Pomej K, Bauer D, Thaler J, Ay C, Quehenberger P, Fritzer-Szekeres M, Peck-Radosavljevic M, Trauner M, Reiberger T, Ferlitsch A; Vienna Hepatic Hemodynamic Lab. Von Willebrand factor indicates bacterial translocation, inflammation, and procoagulant imbalance and predicts complications independently of portal hypertension severity. Aliment Pharmacol Ther. 2018 Apr;47(7):980-988. doi: 10.1111/apt.14522. Epub 2018 Jan 29. PMID 29377193
- [Result] Mandorfer M, Hernandez-Gea V, Garcia-Pagan JC, Reiberger T. Noninvasive Diagnostics for Portal Hypertension: A Comprehensive Review. Semin Liver Dis. 2020 Aug;40(3):240-255. doi: 10.1055/s-0040-1708806. Epub 2020 Jun 18. PMID 32557480
- [Result] Carnevale R, Raparelli V, Nocella C, Bartimoccia S, Novo M, Severino A, De Falco E, Cammisotto V, Pasquale C, Crescioli C, Scavalli AS, Riggio O, Basili S, Violi F. Gut-derived endotoxin stimulates factor VIII secretion from endothelial cells. Implications for hypercoagulability in cirrhosis. J Hepatol. 2017 Nov;67(5):950-956. doi: 10.1016/j.jhep.2017.07.002. Epub 2017 Jul 14. PMID 28716745
- [Result] Ferro D, Quintarelli C, Lattuada A, Leo R, Alessandroni M, Mannucci PM, Violi F. High plasma levels of von Willebrand factor as a marker of endothelial perturbation in cirrhosis: relationship to endotoxemia. Hepatology. 1996 Jun;23(6):1377-83. doi: 10.1002/hep.510230613. PMID 8675154
- [Result] van der Vorm LN, Remijn JA, de Laat B, Huskens D. Effects of Plasmin on von Willebrand Factor and Platelets: A Narrative Review. TH Open. 2018 Jun 7;2(2):e218-e228. doi: 10.1055/s-0038-1660505. eCollection 2018 Apr. PMID 31249945
- [Result] Garcia-Pagan JC, Gracia-Sancho J, Bosch J. Functional aspects on the pathophysiology of portal hypertension in cirrhosis. J Hepatol. 2012 Aug;57(2):458-61. doi: 10.1016/j.jhep.2012.03.007. Epub 2012 Apr 12. No abstract available. PMID 22504334
- [Result] Mandorfer M, Simbrunner B. Prevention of First Decompensation in Advanced Chronic Liver Disease. Clin Liver Dis. 2021 May;25(2):291-310. doi: 10.1016/j.cld.2021.01.003. Epub 2021 Mar 10. PMID 33838851
- [Result] Yilmaz VT, Dincer D, Avci AB, Cetinkaya R. Significant Association between Serum Levels of Von Willebrand Factor (vWF) Antigen with Stages of Cirrhosis. Eurasian J Med. 2015 Feb;47(1):21-5. doi: 10.5152/eajm.2014.0016. PMID 25745341